CLINICAL TRIAL: NCT03971305
Title: A Prospective Multicenters Clinical Cohort Study of the Efficacy and Safety of Stratified Risk Factors for Treatment of Chinese Children With Systemic ALK-positive Anaplastic Large Cell Lymphoma
Brief Title: A Prospective Multicenters Clinical Cohort Study of Stratified Treatment of Chinese Children With Systemic ALK(+) ALCL
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Xiao-Fei Sun, professor, Sun Yat-sen University
Other Study IDs: SCCCG-ALCL-2017-001
Record Dates: First submitted 2019-05-30; First posted 2019-06-03 (Actual); Last update posted 2022-05-09 (Actual); Status verified 2022-05

CONDITIONS: MRD; MDD; Lymphoma, Nonhodgkin; Anaplastic Lymphoma; Pediatric Cancer
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
With the development of molecular biology and precise medical treatment, new challenges have been raised in the diagnosis and treatment of non-Hodgkin lymphoma (NHL) in children. In recent years, the criteria for clinical staging and efficacy evaluation of NHL in children have been updated. Studies in Germany and the United States have shown that pathological types of systemic anaplastic large cell lymphoma (ALCL) in children and adolescents, minimal disseminated disease (MDD) in peripheral blood or bone marrow and minimal residual disease (MRD) are significantly associated with prognosis, suggesting that these factors need to be combined in risk stratification of ALCL patients. Recent studies have also suggested that PET/CT is helpful in evaluating residual lesions in patients with lymphoma after chemotherapy. In order to keep pace with the times in the diagnosis, clinical staging, risk stratification, efficacy evaluation and treatment of NHL in children. We adjusted the original NHL-BFM-90/95 regimen, mainly in the aspects of clinical staging, efficacy evaluation, risk stratification and treatment regimen，etc.

DETAILED DESCRIPTION:
Research purpose:

1. To study the efficacy and safety of SCCCG-ALCL-2017 regimen in children with systemic ALK-positive anaplastic large cell lymphoma.
2. To explore the correlation between MDD or MRD in peripheral blood or bone marrow and the treat response and survival.
3. To explore the feasibility of risk stratification combined with adverse pathological types, dangerous organ invasion and MDD.
4. To investigate the effect of vinblastine maintenance chemotherapy on survival of patients with MRD-positive in peripheral blood after treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Age < 18 years old
2. Pathologically confirmed systemic ALK-positive anaplastic large cell lymphoma
3. Newly diagnosed patients
4. Informed consent of guardian of children patients

Exclusion Criteria:

1. Secondary immunodeficiency disease
2. Second neoplasm
3. Primary cutaneous anaplastic large cell lymphoma
4. Recurrent and progressive patients.

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Systemic ALK-positive anaplastic large cell lymphoma patients # age at diagnosis < 18 years.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2017-05-05 (Actual); Primary Completion 2022-05-05 (Estimated); Study Completion 2025-05-05 (Estimated)

PRIMARY OUTCOMES:
Event-free survival (EFS) | through study completion, maximal eight years
  EFS is defined as time from start of treatment/randomization up to event or to date of last contact for patients without event. The following occurrences are defined as an event: non-response, progressive disease or relapse, treatment related death, death of any other cause or diagnosis of secondary malignancies

SECONDARY OUTCOMES:
Overall survival (OS) | through study completion, maximal eight years
  OS is defined as time from start of treatment/randomization up to death of any
Relapse-free survival (RFS) | through study completion, maximal eight years
  RFS is defined as time from start of treatment/randomization up to event or to date of last contact for patients without event. The following occurrences are defined as an event: non-response, progressive disease, or relapse.
Response rate (RR) | on an average 3 weeks after finish of treatment
  Complete response, partial remission, objective effect, stable disease or progressive disease
Adverse event rate | from the first day of protocol defined treatment until two years after start of protocol defined treatment
  Rate of patients with acute toxicity defined as grade III/IV/V AE

CONTACTS AND LOCATIONS:
Overall Officials: Sun Xiaofei, Study Director — Sun Yat-sen University
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Burkhardt B, Zimmermann M, Oschlies I, Niggli F, Mann G, Parwaresch R, Riehm H, Schrappe M, Reiter A; BFM Group. The impact of age and gender on biology, clinical features and treatment outcome of non-Hodgkin lymphoma in childhood and adolescence. Br J Haematol. 2005 Oct;131(1):39-49. doi: 10.1111/j.1365-2141.2005.05735.x. PMID 16173961
- [Result] Lamant L, McCarthy K, d'Amore E, Klapper W, Nakagawa A, Fraga M, Maldyk J, Simonitsch-Klupp I, Oschlies I, Delsol G, Mauguen A, Brugieres L, Le Deley MC. Prognostic impact of morphologic and phenotypic features of childhood ALK-positive anaplastic large-cell lymphoma: results of the ALCL99 study. J Clin Oncol. 2011 Dec 10;29(35):4669-76. doi: 10.1200/JCO.2011.36.5411. Epub 2011 Nov 14. PMID 22084369
- [Result] Damm-Welk C, Mussolin L, Zimmermann M, Pillon M, Klapper W, Oschlies I, d'Amore ES, Reiter A, Woessmann W, Rosolen A. Early assessment of minimal residual disease identifies patients at very high relapse risk in NPM-ALK-positive anaplastic large-cell lymphoma. Blood. 2014 Jan 16;123(3):334-7. doi: 10.1182/blood-2013-09-526202. Epub 2013 Dec 2. PMID 24297868
- [Result] Sun X, Zhen Z, Lin S, Zhu J, Wang J, Lu S, Chen Y, Zhang F, Sun F, Li P. Treatment outcome of Chinese children with anaplastic large cell lymphoma by using a modified B-NHL-BFM-90 protocol. Pediatr Hematol Oncol. 2014 Sep;31(6):518-27. doi: 10.3109/08880018.2014.939793. Epub 2014 Aug 12. PMID 25116372
- [Result] Le Deley MC, Rosolen A, Williams DM, Horibe K, Wrobel G, Attarbaschi A, Zsiros J, Uyttebroeck A, Marky IM, Lamant L, Woessmann W, Pillon M, Hobson R, Mauguen A, Reiter A, Brugieres L. Vinblastine in children and adolescents with high-risk anaplastic large-cell lymphoma: results of the randomized ALCL99-vinblastine trial. J Clin Oncol. 2010 Sep 1;28(25):3987-93. doi: 10.1200/JCO.2010.28.5999. Epub 2010 Aug 2. PMID 20679620
- [Derived] Chen T, Zeng C, Wang J, Sun F, Huang J, Zhu J, Lu S, Liao N, Zhang X, Chen Z, Yuan X, Yang Z, Guo H, Yang L, Wen C, Zhang W, Li Y, Luo X, Wu Z, Yang L, Liu R, Zheng M, He X, Sun X, Zhen Z. Stratified Treatment in Pediatric Anaplastic Large Cell Lymphoma: Result of a Prospective Open-Label Multiple-Institution Study. Cancer Res Treat. 2024 Oct;56(4):1252-1261. doi: 10.4143/crt.2024.104. Epub 2024 May 28. PMID 38810968